CLINICAL TRIAL: NCT00108615
Title: Effects of Insulin Sensitizers in Subjects With Impaired Glucose Tolerance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Kern, Philip - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CLIN-013-0S3
Record Dates: First submitted 2005-04-15; First posted 2005-04-18 (Estimated); Last update posted 2008-04-25 (Estimated); Status verified 2008-04

CONDITIONS: Glucose Metabolism Disorders; Diabetes
MeSH Terms: conditions — Glucose Metabolism Disorders; Diabetes Mellitus | interventions — Metformin; Pioglitazone; Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): pioglitazone
  Interventions: Drug: Metformin; Drug: Pioglitazone; Radiation: CT scans; Procedure: Oral glucose tolerance test
- 2 (Active Comparator): metformin
  Interventions: Drug: Metformin; Drug: Pioglitazone; Radiation: CT scans; Procedure: Oral glucose tolerance test

INTERVENTIONS:
Drug: Metformin
  Arms: 1
Drug: Pioglitazone
  Arms: 1
Drug: Metformin
  Arms: 2
Drug: Pioglitazone
  Arms: 2
Radiation: CT scans — To measure changes in adipose tissue volumes
Procedure: Oral glucose tolerance test — To detect a change in glucose tolerance

SUMMARY:
Subjects with impaired glucose tolerance will be randomized to receive pioglitazone or metformin for 10 weeks. Measurements of insulin sensitivity, body composition, glucose tolerance, and muscle lipid accumulation will be performed. Adipose tissue and muscle biopsies are performed. The goal of the study is to determine whether the lipotoxiciy of impaired glucose tolerance is ameliorated by pioglitazone.

DETAILED DESCRIPTION:
The progression to type 2 diabetes represents an evolution, which results from a vicious cycle where both glucotoxicity and lipotoxicity act to reduce insulin secretion and insulin action. Lipotoxicity is a new concept, which refers to overaccumulation of lipids in non-adipose tissue reflecting increased free fatty acid delivery. Increased fat content of skeletal muscle and islet cell is associated with insulin resistance and impaired pancreatic -cell function respectively in animal models. Whether lipotoxicity is the link between obesity and diabetes, in humans, and whether reducing intracellular fat content will improve insulin secretion and sensitivity in humans is not known. In this study, we will focus on obese subjects with impaired glucose tolerance (IGT) who have not yet developed glucose toxicity. We will examine insulin secretion, insulin action, hepatic glucose production, and muscle lipid metabolism in response to two insulin sensitizers with two different modes of action. We propose that thiazolidinediones will improve cell function by reversing lipotoxicity as reflective in reduced muscle lipid accumulation.

Hypothesis 1. In subjects with impaired glucose tolerance, who are insulin resistant and also have an insulin secretory defect, thiazolidinediones, but not biguanides, improve cell function.

Hypothesis 2. In subjects with impaired glucose tolerance, thiazolidinediones, but not biguanides, decrease the accumulation of fat in non-adipose tissues including muscle, pancreas, liver and myocardium.

Specific Aim 1. Fifty subjects with impaired glucose tolerance will be recruited and randomized to pioglitazone or metformin treatment

Specific Aim 2. cell function will be evaluated by measuring changes in acute insulin response to glucose and non-glucose secretagogues in subjects with IGT and it will be compared in response to treatment with pioglitazone versus metformin.

Specific Aim 3. The muscle fat content will be evaluated as the surrogate measure for lipotoxicity and overaccumulation of fat in non-adipose tissue. From the muscle biopsy specimens, we will measure the amount of intramyocellular triglyceride before and after treatment with pioglitazone versus metformin.

Specific Aim 4. Adipose tissue cytokine expression is associated with changes in muscle lipid accumulation.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose tolerance
* Body mass index (BMI) of 28-38

Exclusion Criteria:

* Heart disease
* Renal disease
* Liver disease

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-01; Primary Completion 2007-04 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Effects of pioglitazone and metformin on ectopic lipid accumulation | 4 yr

SECONDARY OUTCOMES:
Effects of pioglitazone and metformin on beta cell responsiveness | 4 yr

CONTACTS AND LOCATIONS:
Overall Officials: Philip A Kern, MD, Principal Investigator — Central Arkansas Veterans HCS
Locations (1):
- Central Arkansas Veterans HCS, Little Rock, Arkansas, United States

REFERENCES:
- [Result] Rasouli N, Raue U, Miles LM, Lu T, Di Gregorio GB, Elbein SC, Kern PA. Pioglitazone improves insulin sensitivity through reduction in muscle lipid and redistribution of lipid into adipose tissue. Am J Physiol Endocrinol Metab. 2005 May;288(5):E930-4. doi: 10.1152/ajpendo.00522.2004. Epub 2005 Jan 4. PMID 15632102
- [Result] Di Gregorio GB, Yao-Borengasser A, Rasouli N, Varma V, Lu T, Miles LM, Ranganathan G, Peterson CA, McGehee RE, Kern PA. Expression of CD68 and macrophage chemoattractant protein-1 genes in human adipose and muscle tissues: association with cytokine expression, insulin resistance, and reduction by pioglitazone. Diabetes. 2005 Aug;54(8):2305-13. doi: 10.2337/diabetes.54.8.2305. PMID 16046295
- [Result] Bodles AM, Varma V, Yao-Borengasser A, Phanavanh B, Peterson CA, McGehee RE Jr, Rasouli N, Wabitsch M, Kern PA. Pioglitazone induces apoptosis of macrophages in human adipose tissue. J Lipid Res. 2006 Sep;47(9):2080-8. doi: 10.1194/jlr.M600235-JLR200. Epub 2006 Jun 23. PMID 16799131
- [Result] Yue L, Rasouli N, Ranganathan G, Kern PA, Mazzone T. Divergent effects of peroxisome proliferator-activated receptor gamma agonists and tumor necrosis factor alpha on adipocyte ApoE expression. J Biol Chem. 2004 Nov 12;279(46):47626-32. doi: 10.1074/jbc.M408461200. Epub 2004 Aug 31. PMID 15339912
- [Result] Rasouli N, Yao-Borengasser A, Miles LM, Elbein SC, Kern PA. Increased plasma adiponectin in response to pioglitazone does not result from increased gene expression. Am J Physiol Endocrinol Metab. 2006 Jan;290(1):E42-E46. doi: 10.1152/ajpendo.00240.2005. Epub 2005 Aug 23. PMID 16118250
- [Result] Bodles AM, Banga A, Rasouli N, Ono F, Kern PA, Owens RJ. Pioglitazone increases secretion of high-molecular-weight adiponectin from adipocytes. Am J Physiol Endocrinol Metab. 2006 Nov;291(5):E1100-5. doi: 10.1152/ajpendo.00187.2006. Epub 2006 Jun 27. PMID 16803857
- [Result] Ranganathan G, Unal R, Pokrovskaya I, Yao-Borengasser A, Phanavanh B, Lecka-Czernik B, Rasouli N, Kern PA. The lipogenic enzymes DGAT1, FAS, and LPL in adipose tissue: effects of obesity, insulin resistance, and TZD treatment. J Lipid Res. 2006 Nov;47(11):2444-50. doi: 10.1194/jlr.M600248-JLR200. Epub 2006 Aug 7. PMID 16894240
- [Result] Rasouli N, Kern PA, Reece EA, Elbein SC. Effects of pioglitazone and metformin on beta-cell function in nondiabetic subjects at high risk for type 2 diabetes. Am J Physiol Endocrinol Metab. 2007 Jan;292(1):E359-65. doi: 10.1152/ajpendo.00221.2006. Epub 2006 Sep 12. PMID 16968813
- [Result] Yao-Borengasser A, Rasouli N, Varma V, Miles LM, Phanavanh B, Starks TN, Phan J, Spencer HJ 3rd, McGehee RE Jr, Reue K, Kern PA. Lipin expression is attenuated in adipose tissue of insulin-resistant human subjects and increases with peroxisome proliferator-activated receptor gamma activation. Diabetes. 2006 Oct;55(10):2811-8. doi: 10.2337/db05-1688. PMID 17003347
- [Result] Varma V, Yao-Borengasser A, Rasouli N, Bodles AM, Phanavanh B, Lee MJ, Starks T, Kern LM, Spencer HJ 3rd, McGehee RE Jr, Fried SK, Kern PA. Human visfatin expression: relationship to insulin sensitivity, intramyocellular lipids, and inflammation. J Clin Endocrinol Metab. 2007 Feb;92(2):666-72. doi: 10.1210/jc.2006-1303. Epub 2006 Nov 7. PMID 17090638
- [Result] Wolins NE, Quaynor BK, Skinner JR, Tzekov A, Croce MA, Gropler MC, Varma V, Yao-Borengasser A, Rasouli N, Kern PA, Finck BN, Bickel PE. OXPAT/PAT-1 is a PPAR-induced lipid droplet protein that promotes fatty acid utilization. Diabetes. 2006 Dec;55(12):3418-28. doi: 10.2337/db06-0399. PMID 17130488
- [Result] Yao-Borengasser A, Varma V, Bodles AM, Rasouli N, Phanavanh B, Lee MJ, Starks T, Kern LM, Spencer HJ 3rd, Rashidi AA, McGehee RE Jr, Fried SK, Kern PA. Retinol binding protein 4 expression in humans: relationship to insulin resistance, inflammation, and response to pioglitazone. J Clin Endocrinol Metab. 2007 Jul;92(7):2590-7. doi: 10.1210/jc.2006-0816. Epub 2007 Jun 26. PMID 17595259
- [Result] Varma V, Yao-Borengasser A, Bodles AM, Rasouli N, Phanavanh B, Nolen GT, Kern EM, Nagarajan R, Spencer HJ 3rd, Lee MJ, Fried SK, McGehee RE Jr, Peterson CA, Kern PA. Thrombospondin-1 is an adipokine associated with obesity, adipose inflammation, and insulin resistance. Diabetes. 2008 Feb;57(2):432-9. doi: 10.2337/db07-0840. Epub 2007 Dec 5. PMID 18057090